CLINICAL TRIAL: NCT00328549
Title: A Study to Evaluate the Erythropoietic Response in Hepatitis C Virus (HCV) Patients Receiving Combination Ribavirin (RBV)/Interferon (IFN) Therapy or RBV/PEG IFN
Brief Title: A Study to Evaluate the Erythropoietic Response in Hepatitis C Virus (HCV) Patients Receiving Combination Ribavirin (RBV)/Interferon (IFN) Therapy or RBV/PEG IFN (NATURAL HISTORY-HCV)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ortho Biotech Products, L.P. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR005116
Record Dates: First submitted 2006-05-19; First posted 2006-05-22 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2010-04

CONDITIONS: Hepatitis C; Anemia
Keywords: Natural History,; Hepatitis C Infection; Ribavirin; Pegylated Interferon; Interferon
MeSH Terms: conditions — Hepatitis C; Anemia | interventions — Ribavirin

INTERVENTIONS:
Drug: Pegylated Interferon and Ribavirin

SUMMARY:
The purpose of this study was to describe the time course and extent of hemoglobin (Hb) changes and the erythropoietic response to PEG-IFN/RBV-induced anemia In HCV-infected subjects.

DETAILED DESCRIPTION:
Patients receiving combination therapy for chronic hepatitis C virus (HCV) infection (standard or pegylated interferon alfa [PEG-IFN] in combination with ribavirin [RBV]) frequently develop moderate to severe anemia. In large, prospective, clinical trials of PEG-IFN alfa-2b and PEG-IFN alfa-2a, the reported mean decreases in hemoglobin (Hb) were 2.5 g/dL and 3.7 g/dL, respectively. Furthermore, in a retrospective study, 54% of standard interferon/RBV-treated patients had hemoglobin (Hb) decreases of at least 3 g/dL. It is important to understand the causes, natural history, and risk factors associated with HCV therapy-induced anemia, because such decreases in Hb can result in RBV dose reduction or discontinuation, which may adversely affect the likelihood of a virologic response. Erythropoietin is an endogenous hormone that acts in the bone marrow to increase the number of erythroid progenitor cells. Normally, a decrease in the Hb level is accompanied by an increase in the serum erythropoietin (sEPO) level, which will ultimately normalize the Hb level. The relationship between Hb and sEPO is less apparent in patients with chronic diseases such as cancer and human immunodeficiency virus (HIV) infection. It is not known whether HCV-infected patients receiving combination PEG-IFN/RBV therapy have a similarly diminished erythropoietic response to anemia.

One hundred HCV-infected patients who are receiving combination RBV/IFN or RBV/PEG-IFN therapy will be enrolled in this multicenter study. No study medication will be administered during this study. Weekly blood samples will be collected at specified times during the initial 8 weeks of RBV/IFN or RBV/PEG-IFN therapy. Assessment of laboratory tests, vital signs, incidence and severity of adverse experiences will be obtained.

The objective of this study is to document the pattern of hemoglobin changes and erythropoietic response (from baseline to final assessment, up to Week 8) in HCV-infected patients receiving combination therapy with RBV/IFN or RBV/PEG-IFN. N/A

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent
* HCV- infected patients confirmed by PCR or branched DNA (b-DNA)
* Scheduled to commence combination RBV/IFN or RBV/PEG-IFN therapy on Day 1
* Normal serum creatinine
* Life expectancy > 6 months

Exclusion Criteria:

* HIV-infected patients
* History of any primary hematologic disease
* Anemia attributable to factors such as iron or folate deficiency, pre-treatment
* hemolysis or gastrointestinal bleeding
* Has suspected or confirmed significant hepatic disease from an etiology other than
* HCV (e.g. alcohol, HBV, autoimmune disease etc)
* Current, active substance abuser
* Pregnant or breast feeding
* Women of childbearing potential not taking adequate birth control measures
* Exposure to Epoetin alfa within three (3) months prior to study enrollment or during study
* Transfusion within three (3) months prior to study entry

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2001-10; Study Completion 2002-12 (Actual)

PRIMARY OUTCOMES:
Primary endpoints were change in Hb and sEPO from baseline to week 8 (or early withdrawal)

SECONDARY OUTCOMES:
Other endpoints measured were changes in reticulocytes, platelets, total bilirubin, and RBV dose from baseline to week 8.

CONTACTS AND LOCATIONS:
Overall Officials: Ortho Biotech Products, L.P. Clinical Trial, Study Director — Ortho Biotech Products, L.P.

REFERENCES:
- [Result] Balan V, Schwartz D, Wu GY, Muir AJ, Ghalib R, Jackson J, Keeffe EB, Rossaro L, Burnett A, Goon BL, Bowers PJ, Leitz GJ; HCV Natural History Study Group. Erythropoietic response to anemia in chronic hepatitis C patients receiving combination pegylated interferon/ribavirin. Am J Gastroenterol. 2005 Feb;100(2):299-307. doi: 10.1111/j.1572-0241.2005.40757.x. PMID 15667486
- See also: A Study to Evaluate the Erythropoietic Response in HCV Patients Receiving Combination Ribavirin/Interferon Therapy or Ribavirin/PEG-Interferon — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=929&filename=CR005116_CSR.pdf